CLINICAL TRIAL: NCT06063707
Title: The Effect of rTEM in the Prognosis and Severity of Sepsis Induced ARDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal Investigator, Southeast University, China
Other Study IDs: 2022ZDSYLL402-P01
Record Dates: First submitted 2023-08-31; First posted 2023-10-02 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Sepsis induced ARDS patients who survived
  Interventions: Other: Taking peripheral blood
- Nonsurvivors: Sepsis induced ARDS patients who not survived
  Interventions: Other: Taking peripheral blood

INTERVENTIONS:
Other: Taking peripheral blood — Taking peripheral blood of no more than 3ml

SUMMARY:
To observe the changes of plasma rTEM levels in patients with sepsis, sepsis induced ARDS, and to explore its clinical significance.

DETAILED DESCRIPTION:
90 patients will be included in this study. Blood samples from these patients in the first day, the third day, were maintained and tested to detect the change of rTEM level. Severity of illness and survival status of every patient were recorded within 28 days. The objective is to observe the changes of plasma rTEM levels in patients with sepsis, sepsis induced ARDS, and to explore its clinical significance.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed as Sepsis 3.0 Patients signing informed consent

Exclusion Criteria:

Pregnant women Patients with tumor、hepatitis、liver cirrhosis、acute myocardial infarction、chronic renal tubular nephritis、interstitial pneumonia、acute pancreatitis、systemic lupus erythenatosus、ulcerative colitis、crohn's disease、HELLP syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study enrolled sepsis patients
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 day
  28day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Principal Investigator — Southeast University

IPD SHARING:
Plan to Share IPD: Undecided